CLINICAL TRIAL: NCT02447848
Title: A Multicenter, Open-Label Trial to Evaluate the Safety and Efficacy of the Sufentanil Sublingual Tablet 30 mcg for the Treatment of Acute Pain in Patients in Emergency Room Setting
Brief Title: Open-Label Safety and Efficacy of the Sufentanil Sublingual Tablet 30 mcg for Acute Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAP302
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-07

CONDITIONS: Moderate-to-severe Acute Pain
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sufentanil sublingual tablet 30 mcg (Experimental): Patients may be administered one tablet every 60 minutes as needed during the study period
  Interventions: Drug: sufentanil sublingual 30 mcg tablet

INTERVENTIONS:
Drug: sufentanil sublingual 30 mcg tablet

SUMMARY:
To evaluate the safety and efficacy of sufentanil tablet (ST) 30 mcg in the management of moderate-to-severe acute pain in patients in an emergency room (ER) setting.

DETAILED DESCRIPTION:
The study is a multicenter, open-label trial, in patients 18 years and older, who present to the ER with moderate-to-severe acute pain due to obvious trauma or injury evident on physical examination.

Upon meeting all entrance criteria, patients will be administered up to four doses of sufentanil 30 mcg and remain in the study for 5 hours for safety and efficacy measurements.

Safety will be monitored via periodic measurement of vital signs and continuous monitoring of oxygen saturation, as well as assessment of adverse events (AEs) and the use of concomitant medications.

Efficacy will be assessed by patient reports of pain intensity (PI) and pain relief. A Six-Item Screener (SIS) will be administered before and 1 hour after study drug administration to measure cognitive impairment. The Patient Global Assessment (PGA) and the Healthcare Professional Global Assessment (HPGA) will assess global satisfaction with the method of pain control.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the ER with moderate-to-severe pain due to obvious trauma or injury evident on physical examination.
* Patients classified as American Society of Anesthesiologists (ASA) class I-III
* Patients who are willing and capable of understanding and cooperating with the requirements of the study.
* Patients able to understand and communicate in English.
* Patients who have provided written informed consent and signed the IRB approved consent form.

Exclusion Criteria:

* Patients who have taken an opioid for more than 30 consecutive days, at a daily dose of more than 15 mg of morphine (or equivalent), within the past 3 months (e.g. more than 3 doses per day of Vicodin®, Norco®, Lortab® with 5 mg hydrocodone per tablet).
* Patients who have used any illicit drugs of abuse, abused prescription medication or alcohol (4 or more drinks per day) within one year before the start of the study.
* Patients with an allergy or hypersensitivity to opioids.
* Patients who are currently taking monoamine oxidase inhibitors (MAOIs) or have taken MAOIs within 14 days of the dose of study drug.
* Patients with current sleep apnea that has been documented by a sleep laboratory study or are on home continuous positive airway pressure (CPAP).
* Female patients who are pregnant (positive pregnancy test) or breastfeeding.
* Patients with a medical condition that, in the Investigator's opinion, could adversely impact the patient's participation or safety, conduct of the study, or interfere with the pain assessments, including chronic pain or active infection.
* Patients who present to the ER using supplemental oxygen.
* Patients who have participated in a clinical trial of an investigational drug or device within 30 days of enrollment.
* Patients who are active or reserve duty with the US military.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela P. Palmer, MD, PhD, Study Director — Talphera, Inc
Locations (3):
- United States (3):
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Hermann Memorial Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sufentanil Sublingual Tablet 30 mcg
Started | 76
Completed | 65
Not Completed | 11
Not completed — Patient discharged | 3
Not completed — Lack of Efficacy | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Sufentanil Sublingual Tablet 30 mcg
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 67
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 46

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Summed Pain Intensity Difference (SPID) Over the 1-hour (SPID1).
Description: The primary efficacy endpoint is the time-weighted SPID1 evaluated from the patient questionnaire data. Pain intensity (PI) will be measured using an 11-point numerical rating scale (NRS) with 0 (no pain) and 10 (worst possible pain).
  The patient's rating of PI will be measured at baseline and at 0.25 (15 min), 0.5 (30 min), 0.75 (45 min), 1, 2, 3, 4, and 5 hours following the first dose of study drug.
  The PID at each evaluation time point after the initiation of the first dose is the difference in PI at the specific evaluation time point and baseline pain intensity [PID (evaluation time after the first dose) = PI(baseline) - PI(evaluation time after the first dose)]. The time-weighted SPID1 is the time-weighted summed PID over the 1-hour study period.
  The observed SPID scores ranged from -.70 to 8.00. A negative score indicates an increase in pain intensity and a positive score indicates a decrease in pain intensity.
Time Frame: One hour
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Sufentanil Sublingual Tablet 30 mcg
Number analyzed (Participants) | 76
units on a scale | 2.11 (0.24)

2. Secondary Outcome: TOTPAR1 (Time-weighted)
Description: The total pain relief (TOTPAR) is the time-weighted sum of the pain relief scores over the first hour (15 minutes, 30 minutes, 45 minutes and 1-hour after the first dose of study drug is taken) of the study period.
  The minimum score is 0.00 and the maximum score is 4.00. A higher score indicates greater pain relief.
Time Frame: 1-hour
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Sufentanil Sublingual Tablet 30 mcg
Number analyzed (Participants) | 76
units on a scale | 1.37 (0.12)

3. Secondary Outcome: PI at Each Evaluation Time Point
Description: Pain intensity at each evaluation time point after the first dose of study drug up through 5 hours is evaluated using an 11-point NRS where 0 equals no pain and 10 equals worst possible pain. The score was obtained at Baseline, 15- , 30-, 45- minutes, 1-hour, and 2-hours after the first dose for all patients, and at hours 3, 4, and 5 for cohort 2 (patients 41-76). Scores ranged from 0 -10 for the first two hours, and 2 - 10 for hours three to five.
Time Frame: 5 hours
Population: The first cohort of patients (N=40) received one dose of study drug and the study was completed at two hours. The second cohort of patients (N=36) had the option of remaining in the study through five hours; most patients discontinued the study at 2 hours.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Sufentanil Sublingual Tablet 30 mcg
Number analyzed (Participants) | 76
units on a scale
  Baseline | 8.08 (0.20)
  15-minutes | 6.00 (0.27)
  30-minutes | 6.23 (0.30)
  45-minutes | 5.51 (0.35)
  1-hour | 5.2 (0.36)
  2-hours: number analyzed (Participants) | 68
  2-hours | 5.49 (0.37)
  3-hours: number analyzed (Participants) | 6
  3-hours | 6.83 (1.17)
  4-hours: number analyzed (Participants) | 3
  4-hours | 4.67 (1.20)
  5-hours: number analyzed (Participants) | 1
  5-hours | 2

ADVERSE EVENTS:
Time Frame: For the duration of the patients' participation in the study (while in ER).
Arm/Group | Sufentanil Sublingual Tablet 30 mcg
Serious Adverse Events (participants affected / at risk) | 1/76
Other Adverse Events (participants affected / at risk) | 12/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sufentanil Sublingual Tablet 30 mcg (N=76)
Angina Pectoris (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sufentanil Sublingual Tablet 30 mcg (N=76)
Nausea (Gastrointestinal disorders) | 5 — Adverse events reported in this list are possibly or probably related to study drug
Vomiting (Gastrointestinal disorders) | 3
Oxygen saturation decreased (Investigations) | 2
Somnolence (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other